CLINICAL TRIAL: NCT02244944
Title: The Effect of Ezetimibe-Ursodiol Combination Therapy on Biomarkers of Liver Function and Sterol Balance in Subjects With NAFLD
Brief Title: Ezetimibe-Ursodiol Combination Therapy on Biomarkers of Liver Function and Sterol Balance in Subjects With NAFLD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: Gregory Graf, PhD (Other)
Responsible Party: Sponsor-Investigator, Gregory Graf, PhD, PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-0972-F1V
Record Dates: First submitted 2014-09-10; First posted 2014-09-19 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2018-01

CONDITIONS: Nonalcoholic Fatty Liver Disease (NAFLD)
Keywords: nonalcoholic fatty liver disease; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Ezetimibe; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EZ-URSO Combination Therapy (Experimental): Ursodiol (URSO Forte) 13-15 mg per kg (250-500 mg b.i.d. or t.i.d depending on body weight) combined with Ezetimibe (Zetia) 10 mg o.p.d.
  Interventions: Drug: EZ-Urso combination therapy

INTERVENTIONS:
Drug: EZ-Urso combination therapy — Ursodiol 13-15 mg per kg per day combined with Ezetimibe (Zetia) 10 mg per day
  Other Names: Ezetimibe (Zetia); Ursoldiol (URSO Forte)

SUMMARY:
The purpose of this research is to gather information on the combination Zetia® (Ezetimibe) and Urso Forte® with respect to sterol balance and their effects on biomarkers of liver function in subjects with nonalcoholic fatty liver disease (NAFLD).

DETAILED DESCRIPTION:
The study will be conducted as a prospective open label trial with pre- and post-treatment measures for all dependent variables. This trial will enroll subjects with a clinical diagnosis of nonalcoholic fatty liver disease (NAFLD) by magnetic resonance imaging (MRI), computed tomography (CT) or ultrasound, including those diagnosed with nonalcoholic steatohepatitis (NASH). Subjects will be consented, blood collected and a MRI conducted on the first visit. Patients will be advised on the proper use of the study drug and given the first three month's supply of the study drug to take home with them. For the remaining three months, study drug will be delivered by US mail along with return packaging for the prior three month's study medication in order to monitor compliance. Patients will be called routinely to encourage compliance, retention, and monitor side effects or adverse events. After six months of study drug administration, subjects will return for a follow-up visit. Blood will be drawn, an MRI will be obtained and a post-study questionnaire will be administered.

Duration of Patient Enrollment: 6 months Duration of Study: 18 months

ELIGIBILITY:
Inclusion Criteria:

* Steatosis
* ALT >1.5 times normal
* ALT/AST ratio >1.0
* Normal Kidney Function

Exclusion Criteria:

* Normal ALT within last 6 months
* Advanced fibrosis based on 1) biopsy, if available (Stage 3 or 4 NAFLD), 2) imaging, or 3) lab (platelet count <150,000)
* Daily alcohol use above 20 g/day for women and 30 g/day for men
* Prescription use of ursodiol, ezetimibe, vitamin E, fish oils, thiazolidinediones, insulin, sulfonylureas, HMG-CoA reductase inhibitors
* Weight loss greater than 15% in past 12 months
* Pregnant or breastfeeding
* Body Mass index greater than 50
* Largest body circumference greater than 160 cm
* Claustrophobia
* Allergy to ezetimibe or ursodiol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Graf, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EZ-URSO Combination Therapy
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Study Terminated | 1

BASELINE CHARACTERISTICS:
Arm/Group | EZ-URSO Combination Therapy
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43.5 [33 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Serum Alanine Transaminase (ALT)
Description: Determine if Ezetimibe-Ursodiol combination therapy improves liver function tests (ALT)
Time Frame: 6 months
Population: The trial was terminated early. No data was collected to analyze the primary outcome measure.
Arm/Group | EZ-URSO Combination Therapy
Number analyzed (Participants) | 0

2. Secondary Outcome: Increase in Plasma Lathosterol
Description: Determine if Ezetimibe-Ursodiol combination therapy promotes a net-negative sterol balance as evidenced by an increase in the cholesterol synthesis intermediate, lathosterol, in plasma.
Time Frame: 6 months
Population: The trial was terminated early. No data was collected to analyze the secondary outcome measure.
Arm/Group | EZ-URSO Combination Therapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Reduction in Hepatic Fat Fraction
Description: Determine if Ezetimibe-Ursodiol combination therapy reduces total fat in the liver as assessed by MRI
Time Frame: 6 months
Population: The trial was terminated early. No data was collected to analyze the primary outcome measure.
Arm/Group | EZ-URSO Combination Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | EZ-URSO Combination Therapy
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EZ-URSO Combination Therapy (N=2)
diarrhea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes